CLINICAL TRIAL: NCT00148785
Title: Pharmacokinetics of an Indinavir, Ritonavir and Amprenavir Regimen in HIV-Infected Individuals: A Pilot Study
Brief Title: A Pharmacokinetic (PK) Study of a Combination of Indinavir, Ritonavir, and Amprenavir
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Ighovwerha Ofotokun, Principal Investigator, Emory University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00006856; 04008; 2804G (Other: Other)
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2013-11

CONDITIONS: HIV Infections
Keywords: Antiretroviral drugs; Pharmacokinetic; Indinavir; Ritonavir; Fosamprenavir
MeSH Terms: conditions — HIV Infections | interventions — Indinavir

INTERVENTIONS:
Drug: Indinavir/Ritonavir/Fosamprenavir

SUMMARY:
When individuals who are infected with HIV are started on treatment with HIV medications, the effect of these drugs only lasts for a limited period of time, often because of development of drug resistance by the HIV virus. When this happens, such patients have to be switched to different combinations of HIV medications. However, since the availability of new HIV drugs that are active against resistant virus is limited, HIV care providers are resorting to curtail medications that contain three or more protease inhibitors (PIs). The reason for this is Norvir (ritonavir), a PI that has the ability to boost or increase the blood levels of other PIs in a way that can sometimes overcome the resistance of HIV virus. In addition, it may be more difficult for the virus to overcome two or more drugs with high blood levels, than it is to overcome just one. For these reasons, many clinicians are now using Norvir in combination with two other PIs, including Crixivan (indinavir) plus Lexiva (fosamprenavir), for treating patients who have been exposed to many other HIV medications.

While this may be the case, researchers also know that when two or more PIs are combined, the effects each drug may have on the blood level of other drugs could be different. For example, researchers know from some recent studies that the combination of Norvir, Lexiva, and Kaletra, another PI, leads to an unacceptably low level of both Kaletra and Lexiva. Because researchers can not always assume that when multiple HIV medications are combined, the levels will remain high enough to be effective, the investigators think it will always be reasonable that, before any combination of drugs are used on HIV-infected patients, the effect a combination has on the levels of each of the drugs in the combination should be investigated.

AIMS: The aim of this pilot study therefore is to examine the blood levels of Crixivan, Lexiva, and Norvir when these three drugs are used together as part of a combination treatment for HIV infection.

METHODS: Fifteen (15) HIV-infected volunteers already being treated with a Crixivan and Norvir containing regimen will be recruited from the Grady Infectious Disease Clinic (IDP). Lexiva will be added to this regimen for 5 days, at the end of which participants will be admitted to the Grady General Clinical Research Center (GCRC) where blood samples will be collected at 9 different time points over 12 hours for measurement of blood drug levels.

Pharmacokinetic Analysis: The blood concentrations of Crixivan, Lexiva, and Norvir will be measured by a special technique known as reverse-phase high-performance liquid chromatography with ultraviolet detection.

Statistical Analysis: The blood level information will be summarized by a statistical method. The researchers will then compare the levels of Lexiva in this combination with historically published levels of Lexiva in a study of Lexiva plus Norvir; and that of Crixivan in a study of Crixivan plus Norvir. A difference of 30% or more in drug levels between this study and historical reports will be considered a significant difference.

DETAILED DESCRIPTION:
BACKGROUND: Because of their potent antiviral effects, protease inhibitor (PI)-containing antiretroviral regimens (ARV) have become one of the cornerstones of HIV treatment. Success with their use has however been dampened by increasing emergence of resistant viral gene mutation with consequent treatment failure. Since the availability of newer antiviral agents with activity against resistant viral strains are limited, clinicians are increasingly resorting to ritonavir (RTV) enhanced dual PI therapy to treat salvage patients.

In the presence of RTV, the metabolism of concomitantly administered PIs by the cytochrome P450 3A4 (CYP3A4) isoenzyme is inhibited; higher plasma and tissue drug levels are maintained with less variability. The enhanced pharmacokinetics result in prolonged suppression of viral replication including strains with moderate phenotypic resistance leading to improved therapeutic outcomes. RTV enhanced dual PI therapy offers additional advantages as combinations of PIs with different and non-overlapping mutation patterns would be expected to delay emergence of viral resistance, coupled with the notion that the selection of resistance to two or more agents may require a greater number of mutations than that required to overcome a single PI. Furthermore, these combination regimens often result in reduction in pill burden, food restrictions, and may be associated with more tolerable side effect profiles.

For these reasons, RTV enhanced indinavir (IDV) and fos-amprenavir (fos-APV) combinations appear promising for salvage therapy as these two agents are pharmacokinetically enhanced by RTV, and have unique resistant mutation profiles when compared with other PIs. Additionally, since clinically limiting interaction is known to occur between fos-APV and lopinavir/ritonavir (LPV/r), the interactions between IDV, fos-APV, and RTV may be different in a manner that could be clinically beneficial in salvage therapy. Importantly, we will evaluate IDV/fos-APV/RTV at a dose of 800/700/100 mg bid as we anticipate that fos-APV may lower IDV concentrations similarly to lopinavir (LPV), although likely to a lesser extent; such that a dual benefit of enhanced efficacy and improved tolerability could be achieved. The pharmacokinetic profile of this combination regimen therefore merits evaluation to allay concerns of clinically important drug-drug interactions before introduction into clinical practice.

AIMS: The aim of this pilot study therefore is to evaluate the impact of the addition of fos-APV on the pharmacokinetic parameters (plasma trough concentrations (Cmin), the peak concentrations (Cmax), the elimination half-life (t1/2β), and the area under the concentration-time curve (AUC12)) of IDV and RTV at steady state in HIV infected patients.

METHODS: Fifteen HIV-infected subjects already being treated with IDV/RTV containing ARV therapy (800/100 mg bid) will be recruited from the Grady Infectious Disease Clinic (IDP). Initially, blood samples will be collected at time 0, 1, 2, 3, 4, 6, 8, 10, and 12 hours for a baseline 12-hour pharmacokinetics study of RTV and IDV. Fos-APV 700 mg bid will be added to this regimen for 5 days. At the end of which blood samples will be collected at time 0, 1, 2, 3, 4, 6, 8, 10, and 12 hours for IDV, RTV and APV pharmacokinetic parameters.

Pharmacokinetic Analysis: Plasma concentrations of IDV, APV, and RTV will be determined with sensitive and validated reverse-phase high-performance liquid chromatography (HPLC). The Cmax, Cmin, t1/2β, and AUC12 of these PIs will be determined using non-compartmental pharmacokinetic methods.

Statistical Analysis: IDV and RTV pharmacokinetic indices before and after the addition of fos-APV will be compared using a non-parametric two-sided paired t-test.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or more
* Diagnosis of HIV infection or AIDS as previously established by HIV ELISA test and confirmed by Western blot analysis
* Must have been taking and tolerating IDV/RTV 800/100 mg bid as part of an antiretroviral regimen.

Exclusion Criteria:

* Hepatic abnormality: alanine-aminotransferase (ALT), aspartate- aminotransferase (AST) or total bilirubin (TBR) greater than 3x upper limit of normal
* Renal insufficiency: serum creatinine greater than 2 mg/dl
* Co-infection with hepatitis B and/or C viruses
* Pregnant or breastfeeding
* Use of concurrent medications known to affect IDV or APV concentrations significantly (e.g. rifampin, rifabutin, non-nucleoside reverse transcriptase inhibitor [NNRTI], other PIs, St John's Wort, herbal preparations)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2005-07; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
To compare the steady state Cmax, Cmin, AUC0-12h, and the t1/2 of RTV and IDV in HIV-infected patients treated with IDV/RTV 800/100 mg, in the presence and absence of added fos-APV 700 mg twice a day (bid)

SECONDARY OUTCOMES:
To evaluate the Cmax, Cmin, AUC0-12h, and the t1/2 APV in a double boosted PI regimen of IDV/fos-APV/RTV 800/700/100 mg bid as compared to historical results of APV pharmacokinetics in a regimen of APV/RTV 700/100 mg bid

CONTACTS AND LOCATIONS:
Overall Officials: Igho Ofotokun, MD, MSc, Principal Investigator — Emory University
Locations (1):
- Grady Infectious Diseases Program, Atlanta, Georgia, United States